CLINICAL TRIAL: NCT04348461
Title: Two-treatment,Randomized, Controlled, Multicenter Clinical Trial to Assess the Safety and Efficacy of Intravenous Administration of Expanded Allogeneic Adipose Tissue Adult Mesenchymal Stromal Cells in Critically Ill Patients COVID-19
Brief Title: BAttLe Against COVID-19 Using MesenchYmal Stromal Cells
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of financial support
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network); Hospital General Universitario Gregorio Marañon (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); University of Salamanca (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BALMYS-19
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-05

CONDITIONS: COVID; Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients receiving regular respiratory distress treatment
- Treatment (Experimental): Patients receiving two serial doses of allogeneic and expanded adipose tissue-derived mesenchymal stromal cells
  Interventions: Drug: Allogeneic and expanded adipose tissue-derived mesenchymal stromal cells

INTERVENTIONS:
Drug: Allogeneic and expanded adipose tissue-derived mesenchymal stromal cells — Two serial doses of 1.5 million adipose-tissue derived mesenchymal stem cells per kg
  Arms: Treatment

SUMMARY:
The investigational medicinal product consists of expanded allogeneic mesenchymal stromal cells derived from adipose tissue and administered intravenously.

The objective of this project is to evaluate the safety and efficacy of the administration of expanded allogeneic adipose tissue adult mesenchymal stem cells, in patients infected with SARS-COV-2 with COVID-19 type complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Over 18 years.
* Confirmation of SARS-COV-2 infection by RT-PCR in respiratory sample.
* Respiratory failure requiring intubation and connection to mechanical ventilation, secondary to SARS-CoV-2 infection.
* Criteria for acute respiratory distress: acute bilateral alveolar-interstitial infiltrate not compatible with left ventricular failure (demonstrated with ultrasound or hemodynamic parameters), sudden onset, and blood gas compromise with a PaO2 / FiO2 ratio <200 mm-Hg.
* Women of childbearing potential should have a negative urine pregnancy test performed at the time of study enrollment.
* Written or verbal informed consent from the patient, family member or legal representative.

Exclusion Criteria:

* Any other cause of acute respiratory distress not attributable to SARS-Cov-2.
* RT-PCR of SARS-Cov-2 negative.
* Multi-organ failure (more than three organs)
* Severe respiratory failure requiring extracorporeal support (ECMO) Grave Moderate severe COPD requiring chronic home oxygen therapy, need for prior home oxygen therapy for any reason.
* Pregnancy, lactation and women of childbearing age but who do not take effective contraceptive measures.
* Active tumor disease.
* Previous immunosuppressive treatment.
* Allergy or hypersensitivity to the administered products.
* History of deep vein thrombosis or pulmonary embolism in the last 3 years.
* Participation in other clinical trials during the 3 months prior to the initial visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the administration of allogeneic mesenchymal stem cells derived from adipose tissue assessed by Survival Rate) | 28 days
Safety of the administration of allogeneic mesenchymal stem cells derived from adipose tissue assessed by Adverse Event Rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain